CLINICAL TRIAL: NCT05122312
Title: Comparative Study on the Efficacy of OliNano SEAL and Curodont D' Senz in Treatment of Dentin Hypersensitivity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Asmaa Ahmed Mosleh, Principal Investigator, Al-Azhar University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OPDENT A13
Record Dates: First submitted 2021-03-17; First posted 2021-11-16 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Dentin Hypersensitivity
Keywords: OLiNano SEAL; Curodont D'Senz; Dentin Hypersensitivity; Dye penetration; Dentin permeability
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Intervention Model Description: A total of ninety (90) samples were used in the study, for dentin permeability test (dye penetration test) and Scanning Electron Microscopic examination (SEM) which were randomly divided into two main groups; group A1, completely removed smear layer, group A2, partially removed smear layer. Each group was subdivided into three subgroups according to the desensitizing agent applied: OliNano SEAL, Curodont D'Senz and the control group that were left untreated. Seventy (70) hypersensitive teeth in ten patients were enrolled for the current study. The subjective assessment of dentin hypersensitivity was done prior to the application of the desensitizing agent (baseline) then immediately, 2 weeks, 4 weeks and 3 months after application of the tested materials. Patients were informed to rate their perception to tactile, air and cold stimuli by using Verbal Rating Score (VRS) and Visual Analogue Scale (VAS).
Who Masked: Participant, Care Provider
Masking Description: they don't know the type of intervention used
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Totally removed smear layer (Other): Smear layer is completely removed by etchant of phosphoric acid
  Interventions: Drug: Olinanoseal; Drug: Curodont D'senz
- Partially removed smear layer (Other): Smear layer is partially removed by etchant of phosphoric acid
  Interventions: Drug: Olinanoseal; Drug: Curodont D'senz

INTERVENTIONS:
Drug: Olinanoseal — it contains nanometer particles of fluoroapatite and calcium fluoride - guarantees the resistance to cracks and abrasion. At the same time insoluble nano-fluoroapatites fill all enamel microcracks and closes open dentinal tubules.
  Other Names: silicone polymer protector varnish
Drug: Curodont D'senz — This agent contains p 11-4 peptide in addition to fluoride
  Other Names: Self assembling peptide containing desensitizing agent

SUMMARY:
This study was conducted to evaluate and compare the efficacy of Olinanoseal and Curodont D'Senz in treatment of dentin hypersensitivity.

DETAILED DESCRIPTION:
Materials and Methods:- A total of ninety (90) samples were used in the study, for dentin permeability test (dye penetration test) and Scanning Electron Microscopic examination (SEM) which were randomly divided into two main groups; group A1, completely removed smear layer, group A2, partially removed smear layer. Each group was subdivided into three subgroups according to the desensitizing agent applied: OliNano SEAL, Curodont D'Senz and the control group that were left untreated. Seventy (70) hypersensitive teeth in ten patients were enrolled for the current study. The subjective assessment of dentin hypersensitivity was done prior to the application of the desensitizing agent (baseline) then immediately, 2 weeks, 4 weeks and 3 months after application of the tested materials. Patients were informed to rate their perception to tactile, air and cold stimuli by using Verbal Rating Score (VRS) and Visual Analogue Scale (VAS).

ELIGIBILITY:
Inclusion Criteria:

1. Presence of a minimum of four hypersensitive teeth in each patient.
2. Patients with teeth recorded a discomfort score of two or more to tactile, cold and air stimulation.
3. Teeth having hypersensitivity only on the facial aspect.
4. Patients' willingness to participate in the study

Exclusion Criteria:

1. Patients with any medical or dental condition that could impact the study results during its expected length.
2. Patients with a history of drug addictions and use of potent analgesic and/ or anti-inflammatory drugs.
3. Patients who refused to give their consents.
4. Patients with any extensive or unsatisfactory restorations, prosthesis or orthodontic appliances which involve the cervical areas

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2021-01-12 (Actual)

PRIMARY OUTCOMES:
dentin hypersensitivity | 2 minutes
  pain score (visual analogue scale VAS ["minmum =0 {best}, maximum=10 {worst}] and verbal rating scale VRS ["minmum =0 {best}, maximum=4 {worst}])
dentin hypersensitivity | 2 weeks
  pain score (visual analogue scale VAS ["minmum =0 {best}, maximum=10 {worst}] and verbal rating scale VRS ["minmum =0 {best}, maximum=4 {worst}])
dentin hypersensitivity | 4 weeks
  pain score (visual analogue scale VAS ["minmum =0 {best}, maximum=10 {worst}]) and verbal rating scale VRS ["minmum =0 {best}, maximum=4 {worst}])
dentin hypersensitivity | 3 months
  pain score (visual analogue scale VAS ["minmum =0 {best}, maximum=10 {worst}] and verbal rating scale VRS ["minmum =0 {best}, maximum=4 {worst}])

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa A mosleh, lecturer, Study Chair — lecturer, faculty of dental medicine, Al-Azhar university
Locations (1):
- Faculty of dental Medicine for girls, Al-AZhar University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No